CLINICAL TRIAL: NCT02986503
Title: A European Treatment Protocol for Bone-sarcoma in Patients Older Than 40 Years
Brief Title: European Study in Bone Sarcoma Patients Over 40 Years
Acronym: EUROBOSS
Status: Completed | Type: Observational
Sponsor: Italian Sarcoma Group (Network)
Collaborators: Scandinavian Sarcoma Group (Other); Cooperative Osteosarcoma Study Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: EURO-B.O.S.S
Record Dates: First submitted 2016-11-25; First posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Spindle Cell Sarcoma of Bone; Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Doxorubicin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chemotherapy for Good responder: Doxorubicin + cisplatin + ifosfamide Pre-operative and post-operative chemotherapy for patients with good responder high grade osteosarcoma
  Interventions: Drug: Doxorubicin+cisplatin+ifosfamide
- Chemotherapy for Poor responder: Doxorubicin+cisplatin+ifosfamide+methotrexate Pre-operative and post-operative chemotherapy for patients with poor responder high grade osteosarcoma
  Interventions: Drug: Doxorubicin+cisplatin+ifosfamide+methotrexate

INTERVENTIONS:
Drug: Doxorubicin+cisplatin+ifosfamide — Chemotherapy for Good responder high grade osteosarcoma
  Other Names: Doxorubicin,cisplatin,ifosfamide
  Groups: Chemotherapy for Good responder
Drug: Doxorubicin+cisplatin+ifosfamide+methotrexate — Chemotherapy for Poor responder high grade osteosarcoma
  Other Names: Doxorubicin,cisplatin,ifosfamide,methotrexate
  Groups: Chemotherapy for Poor responder

SUMMARY:
The study is a first step of a process to establish the standard chemotherapy treatment with the aim to improve outcome for patients with these rare tumours. For this reason the study will be non-controlled clinical trial.

In this regard, the study aims to determine the feasibility of intensive chemotherapy in this age group, and/or separate efficacy analyses according to the different histologic categories and whether the number of patients recruited by the co-operating groups permits future randomised studies.

DETAILED DESCRIPTION:
Wide surgical removal of the tumor with the addition of a systemic treatment based on the antineoplastic drugs active against osteosarcoma (Adriamycin, Cisplatin, Ifosfamide, Methotrexate). The use of radiation therapy will be given to patients with unresectable tumors. It is recommended in patients who underwent inadequate surgical removal of the tumor. The addition of radiation therapy can not compensate for an adequate surgical treatment.

All the patients eligible for the study will receive the planned systemic treatment. Depending on clinical features, and feasibility of adequate surgical removal of the tumor, patients may receive primary chemotherapy followed by a postoperative chemotherapy treatment or only an adjuvant chemotherapy. In case of immediate surgery, patients will receive an adjuvant treatment with the 3-drug regimen (Cisplatin-Adriamycin-Ifosfamide).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of high-grade sarcoma of bone of any site.
2. Histologic types: osteosarcoma (high-grade surface, central primary and secondary), fibrosarcoma, malignant fibrous histiocytoma, leiomyosarcoma, dedifferentiated chondrosarcoma, angiosarcoma.
3. Age: 41 - 65
4. Normal bone marrow, hepatic, cardiac and renal function
5. Absence of contraindications to the use of cisplatin, adriamycin, and ifosfamide
6. Written informed consent

Exclusion Criteria:

1. Planned chemotherapy and/or follow-up not feasible
2. Previous chemotherapy treatment, which contraindicates the use of one or more drugs, included in the present protocol
3. Previous chemotherapy treatment for the current tumor
4. White blood count < 3.0 x 109/L, and platelets < 100 x 109/L
5. Creatinine clearance < 70 ml/min
6. Left ventricular ejection fraction < 55% or fractional shortening rate of the left ventricle <28%
7. Serum transaminases and bilirubin > 2 times the normal values
8. ECOG performance status > 2
9. Chondrosarcoma or small/round cell bone sarcoma including mesenchymal chondrosarcoma and Ewing's family tumors.

Ages: 41 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 40 years with highly malignant spindle cell sarcoma of bone
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2002-01; Primary Completion 2015-12 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Event-free survival | from the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 168 months.
  Survival without any events related to disease (e.g: progression, relapse or osteosarcoma related death)

SECONDARY OUTCOMES:
Progression-free survival | from the date of randomization until the date of first documented progression of disease, whichever came first, assessed every 6 months, up to 168 months
  Survival without progression of disease
Disease-free survival | from the date of randomization until the date of first documented progression of disease, whichever came first, assessed every 6 months, up to 168 months
  Survival without disease
Metastasis-free survival | from the date of randomization until the date of first documented progression in term of metastasis, whichever came first, assessed every 3 months, up to 168 months
  Survival without metastasis
Overall survival | from the date of randomization until the end of the study, assessed every 3 months, up to 168 month
  Global patients survival evaluation after treatment
Chemotherapy toxicity | Every 3 weeks
  Number and grade of adverse events related to the study treatments

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Ferrari, MD, Principal Investigator — Italian Sarcoma Group
Locations (3):
- Cooperative Osteosarcoma Study Group, Stuttgart, Germany
- Istituti Ortopedici Rizzoli - Unit of Chemotherapy of Muscoloskeletal Tumors, Bologna, Bologna, Italy
- Scandinavian Sarcoma Group, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Anonymized results will be available upon request at the end of the study and public available into the repository systems like Clinicaltrial.gov

REFERENCES:
- See also: Euroboss I - A European treatment protocol for bone sarcoma in patients older than 40 years — http://www.ssg-org.net/wp-content/uploads/2011/05/Euroboss1.pdf